CLINICAL TRIAL: NCT00120432
Title: Single Dose of 1% Tropicamide and 10% Phenylephrine for Pupillary Dilation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Yosanan Yospaiboon, Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE461104
Record Dates: First submitted 2005-07-11; First posted 2005-07-18 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Eye Diseases
Keywords: single dose; mydriatic drug; pupillary dilation
MeSH Terms: conditions — Eye Diseases; Mydriasis | interventions — Tropicamide; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Active Comparator): single dose vs three doses of 1%tropicamide and 10%phenylephrine
  Interventions: Drug: 1% tropicamide and 10% phenylephrine

INTERVENTIONS:
Drug: 1% tropicamide and 10% phenylephrine — single dose vs three doses of 1%tropicamide and 10%phenylephrine

SUMMARY:
The purpose of this study is to compare the efficacy on pupillary dilation between the single dose versus the three doses of 1% tropicamide with 10% phenylephrine for complete ocular examination.

DETAILED DESCRIPTION:
To the best of the authors' knowledge, there have been no clinical trials using an appropriate regimen for pupillary dilation up until now. Therefore, the authors were interested to find out the most appropriate regimen for complete ocular examination, based on the finding that a pupil diameter of 6 mm or greater is adequate for indirect ophthalmoscopy. The authors hypothesize that a single dose of 1% tropicamide and 10% phenylephrine is adequate to complete the job and are conducting this prospective randomized clinical controlled trial to prove the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 80 years old
* dark iris
* require binocular indirect ophthalmoscopy for complete ocular examination
* signed written consent forms

Exclusion Criteria:

* history of ocular trauma
* history of intraocular surgery
* history of laser treatment
* previous eye drop instillation that may affect pupillary dilation
* ocular diseases that may affect pupil size such as Horner's syndrome, Adies' pupil, glaucoma and uveitis
* history of diabetes mellitus, severe hypertension and cardiovascular diseases

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-12; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
horizontal pupil diameter | 30 min

SECONDARY OUTCOMES:
systolic blood pressure | 30 min
diastolic blood pressure | 30 min
heart rate | 30 min
adverse drug reaction | 30 min

CONTACTS AND LOCATIONS:
Overall Officials: Yosanan Yospaiboon, M.D., Principal Investigator — Faculty of Medicine, Khon Kaen University
Locations (1):
- Srinagarind Hospital, Khon Kaen, Changwat Khon Kaen, Thailand

REFERENCES:
- [Result] Ratanapakorn T, Yospaiboon Y, Chaisrisawadsuk N. Single dose of 1% tropicamide and 10% phenylephrine for pupil dilation. J Med Assoc Thai. 2006 Nov;89(11):1934-9. PMID 17205877